CLINICAL TRIAL: NCT02911623
Title: Safety and Feasibility of the Shockwave Lithoplasty® System for the Treatment of Peripheral Vascular Stenosis
Acronym: BTK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shockwave Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TD 0258
Record Dates: First submitted 2016-09-16; First posted 2016-09-22 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lithoplasty Treatment (Experimental): Patients in this group will receive treatment with the Shockwave Lithoplasty® System which uses lithotripsy-enhanced, low-pressure balloon dilation of calcified stenotic peripheral arteries.
  Interventions: Device: Shockwave Lithoplasty® System

INTERVENTIONS:
Device: Shockwave Lithoplasty® System — The Shockwave Lithoplasty® System is a proprietary lithotripsy-enhanced balloon catheter that is designed to be delivered through the peripheral arterial system of the lower extremities to the site of calcified stenosis. Activating the lithotripsy within the device will generate pulsatile mechanical energy within the target treatment site, disrupt calcium within the lesion and allow subsequent dilation of a peripheral artery stenosis using low balloon pressure. The system consists of a balloon catheter with multiple integrated lithotripsy electrodes, and a generator.

SUMMARY:
To observe early safety and performance of the Shockwave Medical Lithoplasty® System (specifically, Lithoplasty® Catheters: 2.5 x 60mm, 2.75 x 60mm, 3.0 x 60mm, 3.25 x 60mm, and 3.5 x 60mm) in subjects to demonstrate that the Shockwave device can safely and effectively deliver localized pulsatile mechanical energy for balloon dilation of calcified, stenotic, infrapopliteal arteries.

DETAILED DESCRIPTION:
Shockwave Medical, Inc. intends to conduct a prospective, single-arm, multi-center, clinical study designed to evaluate the early safety and performance of the Shockwave Lithoplasty® System in subjects with moderate to heavily calcified peripheral arteries with 2.5mm to 3.5mm reference vessel diameter at the target site. The Shockwave Lithoplasty® System is indicated for lithotripsy-enhanced, low-pressure balloon dilation of calcified, stenotic peripheral arteries in patients who are candidates for percutaneous therapy. Up to twenty subjects will be enrolled and treated with Lithoplasty® System.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is able and willing to comply with all assessments in the study.
2. Subject or subject's legal representative have been informed of the nature of the study, agrees to participate and has signed the approved consent form.
3. Age of subject is >18.
4. Rutherford Clinical Category 1 - 5.

Angiographic Inclusion Criteria:

1. Single or multiple target lesion(s) is/are located in a de novo artery distal to the trifurcation vessels and extends to and ends above the ankle
2. Target vessel reference diameter is between 2.5mm and 3.5mm by visual estimate
3. Target lesion with diameter stenosis ≥50% by investigator via visual estimate
4. If inflow disease >50% proximal to the trifurcation vessels is present, and it can be treated with POBA, stent or Lithoplasty and without complications.
5. Target lesion is ≤150mm in length
6. Subject has at least one patent tibial vessel (>50%) with run-off to the foot.
7. No evidence of aneurysm or acute thrombus in target vessel.
8. Any presence of calcification within the target lesion as assessed by imaging (radiograph, CT or angiography).

Exclusion Criteria:

1. Rutherford Clinical Category 6.
2. Target lesion is within only lower extremity vessel with < 50% stenosis.
3. Gangrene of the lower extremity.
4. Planned major amputation of the target leg.
5. Previously implanted stent in the treatment lesion
6. Target lesion length exceeds 150mm.
7. Patient has chronic total occlusion of target lesion.
8. Patient has significant stenosis (>50% stenosis) or occlusion of inflow tract (e.g., iliac or common femoral) not successfully treated with POBA, stent or Lithoplasty and without complications.
9. Patient in whom antiplatelet, anticoagulant, or thrombolytic therapy is contraindicated.
10. Patient has known allergy to contrast agents or medications used to perform endovascular intervention that cannot be adequately pre-treated.
11. Patient has known allergy to urethane, nylon, or silicone.
12. Patient is pregnant or nursing.
13. Patient is participating in another research study involving an investigational agent (pharmaceutical, biologic, or medical device) that has not reached the primary endpoint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Composite of new-onset Major Adverse Events (MAE) | Procedure through 30 days post procedure
  Death Myocardial infarction Need for emergency surgical revascularization of the target limb. Amputation of target limb.
Efficacy | Peri-Procedural
  Acute reduction in percent (%) diameter stenosis of target lesion

SECONDARY OUTCOMES:
Procedural Success | Peri-Procedural
  The ability of the Shockwave Lithoplasty® System to achieve a post-shockwave residual diameter stenosis of ≤50%

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Brodmann, MD, Principal Investigator — Universitätsklinikum LKH Graz
Locations (4):
- Austria (2):
  - Medizinische Universitaet Graz, Graz
  - Hanusch Krankenhaus, Vienna
- Department of Angiology - Universitats Herzzentrum Freiburg, Bad Krozingen, Baden-Wurttemberg, Germany
- Auckland City Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Brodmann M, Holden A, Zeller T. Safety and Feasibility of Intravascular Lithotripsy for Treatment of Below-the-Knee Arterial Stenoses. J Endovasc Ther. 2018 Aug;25(4):499-503. doi: 10.1177/1526602818783989. Epub 2018 Jun 18. PMID 29911480